CLINICAL TRIAL: NCT05684172
Title: Trial of Intra-arterial Tenecteplase Following Successful Endovascular Thrombectomy on Safety and Efficacy in Patients With Large Vessel Occlusion of Posterior Circulation - a Multicenter Randomized Clinical Trial (ATTENTION IA)
Brief Title: Intra-arterial TNK Following Endovascular Thrombectomy in Patients With Large Vessel Occlusion of Posterior Circulation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Wei Hu, Professor, The First Affiliated Hospital of University of Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATTENTION IA
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Acute Ischemic Stroke; Intracranial Artery Occlusion; Endovascular Thrombectomy
Keywords: thrombectomy; endovascular treatment; mechanical thrombectomy techniques; tenecteplase
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endovascular thrombectomy (Active Comparator): For patients randomized to the control group, EVT has to be completed within 24 hours of stroke onset. The choice of EVT strategy will be made by the treating neurointerventionalist. All mechanical thrombectomy devices for EVT, which are approved by CFDA for this purpose, are allowed in the trial.
  Interventions: Other: endovascular thrombectomy alone
- endovascular thrombectomy+intra-arterial tenecteplase (Experimental): For patients randomized to the endovascular treatment arm, tenecteplase will be injected according to protocol, proceeding to inject TNK through a distal access catheter or microcatheter located proximal to the residual thrombus (if still present) and distally to the origin of the lenticulostriates branches. The administration of TNK will be infused for 15 seconds.
  Interventions: Drug: Tenecteplase; Other: endovascular thrombectomy alone

INTERVENTIONS:
Drug: Tenecteplase — If patients are randomized and assigned to receive intra-arterial tenecteplase thrombolysis, tenecteplase will be injected according to protocol, proceeding to inject TNK through a distal access catheter or microcatheter located proximal to the residual thrombus (if still present) and distally to the origin of the pontine arteries.
  Arms: endovascular thrombectomy+intra-arterial tenecteplase
Other: endovascular thrombectomy alone — Patients will receive randomization if the eTICI score on cerebral angiography is 2b-3 and will stop the procedure if they have been assigned to the control group.

SUMMARY:
Rationale: Recently, one prospective multicenter RCT reported a potential beneficial effect of intra-arterial alteplase following successful endovascular thrombectomy (EVT) in patients with an acute intracranial large vessel occlusion. In 2018, another prospective multicenter RCT supported the superiority of tenecteplase over alteplase in ischemic stroke patients with large vessel occlusion.

Objective: To assess the effect of EVT in addition to intra-arterial tenecteplase compared to EVT alone, in patients with large vessel occlusion of posterior circulation, on functional and safety outcomes.

Study design: This is a parallel group, randomized clinical trial of EVT with IA-TNK versus EVT. The trial has observer blind assessment of the primary outcome and of neuro-imaging at baseline and follow-up.

Study population: Patients with acute intracranial large vessel occlusion of posterior circulation and an eTICI 2b-3 after EVT.

Main study parameters/outcomes: The primary effect parameter will be excellent functional status at day 90 defined as a modified Rankin Score (mRS) of 0-1. The estimate will be adjusted for the known prognostic variables age, pre-stroke mRS, time from onset to randomization, stroke severity (NIHSS) and collaterals and adjusted and unadjusted estimates with corresponding 95% confidence intervals will be reported.

ELIGIBILITY:
Inclusion criteria

* Acute ischemic stroke patients with symptomatic intracranial large vessel occlusion (LVO) in the intracranial vertebral artery, basilar artery, or the P1 segment of the posterior cerebral artery.
* Treated with endovascular thrombectomy (EVT) resulting in an eTICI score 2b50/3 at end of the procedure.
* Age of 18 years or older;
* National Institutes of Health Stroke Scale (NIHSS) score on admission≥6;
* Posterior Circulation ASPECTS ≥ 6 on CT/CTA-Source Images/MRI-DWI.
* Time from estimated time of basilar artery occlusion to randomization<24 hours;
* Written informed consent.

Exclusion criteria

* Pre-existing dependency with mRS >1;
* Contraindication to Intravenous Thrombolysis (except time to therapy);
* Complete clinical recovery in the angiography suite by end of EVT procedure;
* Pregnancy; if a woman is of childbearing potential a urine or serum beta HCG test is positive;
* Severe contrast allergy or absolute contraindication to iodinated contrast;
* Participation in other investigational drug or device clinical trials;
* Systolic pressure >185 mmHg or diastolic pressure >110 mmHg, and cannot be controlled by antihypertensive drugs;
* Known genetic or acquired bleeding diathesis, lack of anticoagulant factors, or oral anticoagulant drugs and INR > 1.7, or treated with direct oral anticoagulant agents in the prior 48 hours;
* platelets <100 000/mm3, aPTT >40 s, or PT >15 s; Blood glucose < 2.7 or >22.2 mmol/L;
* Severe renal Failure as defined by a serum creatinine > 3.0 mg/dl (or 265.2 μmol/l) or glomerular Filtration Rate [GFR] < 30, or patient requires hemodialysis or peritoneal dialysis;
* Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT or MRI scan is normal;
* Suspicion of aortic dissection;
* Presumed vasculitis or septic embolization;
* Life expectancy < 1 year;
* Patients that cannot complete 90-day follow-up (e.g. no fixed residence, overseas patients, etc.)；
* CT/MR shows intracranial hemorrhage;
* Ischemic stroke within 3 months;
* Severe head trauma within 3 months;
* Major surgery or severe trauma within the last 2 weeks.
* History of prior intracranial hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
a modified Rankin Score of 0-1 | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)

SECONDARY OUTCOMES:
a modified Rankin Score of 0-3 | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Modified Rankin Score | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
NIHSS score | 24 hours after procedure
  The NIHSS is an ordinal hierarchical scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit.
mortality | 90 (± 14 days) after procedure
  (Number of subjects who died at 90-day follow-up/total number of subjects who participated in 90-day follow-up) x100%
symptomatic intracerebral hemorrhage (ICH) | within 72 hours after procedure
  SICH means any hemorrhage with neurological deterioration, as indicated by an NIHSS score that was higher by ≥4 points than the value at baseline or the lowest value in the first 72 hours or any hemorrhage leading to death.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of USTC, Division of Life Sciences and Medicine, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu W, Nguyen TN, Qureshi M, Chen Z, Tao C, Li R, Yi TY, Feng G, Su J, Cui T, Cao Z, Wang H, Zeng G, Yuan G, Jing X, Luo C, Zhu Y, Qureshi AI, Nogueira RG, Liu X, Abdalkader M. Noncontrast CT vs CT Perfusion Imaging in Patients With Basilar Artery Occlusion: Analysis of the ATTENTION and ATTENTION IA Trials. Neurology. 2025 Aug 12;105(3):e213911. doi: 10.1212/WNL.0000000000213911. Epub 2025 Jul 17. PMID 40674670
- [Derived] Hu W, Tao C, Wang L, Chen Z, Li D, Chen W, Yi T, Xu L, Yu C, Wang T, Yao X, Cui T, Yuan G, Su J, Chen L, Zhou Z, Ma Z, Wang J, Wang B, Han H, Wang H, Chen J, Zhou P, Cao Z, Ren Y, Cai X, Shi H, Zhang G, Yu L, Yuan X, Li J, Zeng G, Ni C, Li T, Wu Y, Li Y, Li K, Liu Y, Wang Y, Jin Y, Liu H, Wen J, Sun J, Zhu Y, Li R, Zhang C, Liu T, Song J, Wang L, Cheng J, Qureshi AI, Nguyen TN, Saver JL, Nogueira RG, Liu X. Intra-arterial tenecteplase after successful endovascular recanalisation in patients with acute posterior circulation arterial occlusion (ATTENTION-IA): multicentre randomised controlled trial. BMJ. 2025 Jan 14;388:e080489. doi: 10.1136/bmj-2024-080489. PMID 39809509
- [Derived] Tao C, Li R, Sun J, Zhu Y, Wang L, Zhang C, Liu T, Song J, Qureshi AI, Abdalkader M, Nguyen TN, Saver JL, Nogueira RG, Hu W. Intra-arterial tenecteplase following endovascular therapy in patients with acute posterior circulation arterial occlusion: study protocol and rationale. J Neurointerv Surg. 2024 Dec 26;17(e1):e68-e73. doi: 10.1136/jnis-2023-021076. PMID 38124230